CLINICAL TRIAL: NCT06023693
Title: A Study on the Effectiveness of a Guided E-health Sleep and Biological Clock Intervention in University Students (i-Sleep & BioClock)
Brief Title: Effectiveness of a Guided Self-help Intervention for Improving Sleep in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Spinhoven, Prof. dr. Philip Spinhoven, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i-Sleep&BioClockRCT
Record Dates: First submitted 2023-08-03; First posted 2023-09-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Insomnia
Keywords: sleep; guided self-help; CBTi; e-health; university students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided online self-help intervention (Experimental): The intervention will be a guided e-health intervention based on CBTi principles (i-Sleep & BioClock). It consists of 5 modules, to be completed in about 5 weeks, and is aimed at improving sleep in university students. The intervention will be entirely held online and will be supported by e-coaches. The topics covered will be sleep hygiene, psychoeducation on sleep and the biological clock, sleep restriction, stimulus control, worrying and relaxation, dysfunctional thoughts, and relapse prevention.
  Interventions: Behavioral: i-Sleep & BioClock
- Online psychoeducation (Active Comparator): The control group will receive access to the platform and to the sleep diary. Their intervention will consist of brief, unstructured online PE for insomnia based on recognized sleep hygiene advice, for example, recommendations about evening routines, and use of alcohol and caffeine. Students will be advised to monitor their sleep in the diary. In contrast to the intervention group, the control group will not receive support of an e-coach. Key differences to the CBTi group are that the online PE (1) does not provide individualized support by an e-coach; (2) includes less content, and (3) is not delivered in a step-by-step manner, but will be provided all at once.
  Interventions: Behavioral: Online Psychoeducation

INTERVENTIONS:
Behavioral: i-Sleep & BioClock — Module 1 Psychoeducation about normal sleep and insomnia, Psychoeducation on the biological clock: the circadian rhythm, chronotypes, zeitgebers, importance of light behaviour Basic sleep hygiene: information about behaviours that are known to promote or impede sleep e.g. performing physical exercise or the use of caffeine Module 2 Sleep restriction and stimulus control: patients are taught to use the bedroom only to sleep and to restrict the time in bed to the average amount of night-time sleep Module 3 Worrying and relaxation: audio files with progressive muscle relaxation exercises are offered and techniques to stop worrying (e.g. thought blocking, evaluation and worry time) Module 4 Erroneous cognitions about sleep: the basics of cognitive behavioural therapy are explained and the most common erroneous ideas about insomnia are discussed Module 5 Summary and plan for the future
  Arms: Guided online self-help intervention
Behavioral: Online Psychoeducation — Online psychoeducation about sleep and the biological clock, basic sleep hygiene
  Arms: Online psychoeducation

SUMMARY:
This randomized controlled trials aims to assess the effectiveness of an online guided self-help intervention ('i-Sleep & BioClock') based on CBTi principles for university students' sleep problems. The study will involve 192 students with subthreshold insomnia who will be randomized to the intervention or online psychoeducation. The intervention consists of 5 modules completed in about 5 weeks, supported by e-coaches. Outcomes include insomnia severity, mental health symptoms, functioning, quality of life, and academic performance, measured at baseline, post-treatment (6 weeks after baseline), and 18 weeks follow-up.

DETAILED DESCRIPTION:
Rationale: University students often suffer from sleep problems which affect their mental health and daily functioning. Cognitive behavioural therapy for insomnia (CBTi) has been proven effective in adults, but research in university students is still limited. The investigators hypothesize that a guided e-health self-help intervention based on CBTi principles ('i-Sleep & BioClock') could offer convenient treatment to students with sleep problems by reducing insomnia severity and improving mental health outcomes.

Objective: The aim of this randomized controlled trial is to assess the effectiveness of a guided e-health sleep and biological clock intervention on sleep, mental health symptoms (depression and anxiety), functioning, quality of life, and academic performance in university students.

Study design: This is a two-arm parallel group superiority randomized controlled trial, comparing a guided e-health intervention based on CBTi to online psychoeducation (PE).

Study population: The aim is to include 192 university students (Bachelor, Master and PhD) with at least subthreshold insomnia (Insomnia Severity Index ≥ 10), aged ≥ 16, who are able to speak Dutch or English, and are affiliated to one of the nine participating universities. Students with current suicidal ideation are excluded.

Intervention: The intervention will be a guided e-health intervention based on CBTi principles (i-Sleep & BioClock). It consists of 5 modules, to be completed in about 5 weeks, and is aimed at improving sleep in university students. The intervention will be entirely held online and will be supported by e-coaches.

Main study parameters/endpoints: The primary outcome will be insomnia severity. Secondary outcomes will be depression, anxiety, daily functioning, academic performance, quality of life, and sleep & light exposure diary outcomes. Outcomes will be measured at baseline, at post-treatment (6 weeks after baseline), and at 18 weeks follow-up. Mediators such as shift in chronotype and light exposure will be examined at baseline, mid-treatment, and post-treatment

ELIGIBILITY:
Inclusion Criteria:

* Being fluent in Dutch and/or English
* Being enrolled as a student (Bachelor, Master or PhD) in one of the Caring Universities partner universities
* Being ≥ 16 years old
* Having self-reported sleep problems; Insomnia Severity Index ≥ 10

Exclusion Criteria:

* Regular night shifts (Not being able to comply to the intervention due to regular night shift, meaning work between 2AM and 6AM at least once a week)
* Current risk for suicidal behaviour

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline (T0), 3 weeks after baseline (T1), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  7-item self-report instrument to assess insomnia severity, scores 0-28, higher scores indicating more insomnia severity

SECONDARY OUTCOMES:
Sleep efficiency (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Sleep onset latency (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Wake after sleep onset (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Early morning awakening (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Total sleep time (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Time spent outside (in minutes) | Change from week 1 to week 7
  Derived from sleep and light exposure diary
Screen use before bed | Change from week 1 to week 7
  Yes/ No question. Derived from sleep and light exposure diary
Munich Chronotype Questionnaire (MCTQ) | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  Self-rated scale to assess individual phase of entrainment on work and work-free days, Addresses questions about: bedtime (actual time), time spent in bed awake before deciding to turn off the lights (in minutes), how long it takes to fall asleep (in minutes), wake up time (actual time), get up time (actual time) on work and work-free days. MCTQ uses the midpoint between sleep on- and offset on free days (mid-sleep on free days, MSF) to assess chronotype. The MCTQ chronotype is expressed in local time, in which earlier time refers to earlier chronotype and later time to later chronotype.
Patient Health Questionnaire (PHQ-9) | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  9-items self-report instrument for severity of depressive symptoms, scores ranging from 0-27, higher scores indicating more severe depression
Generalised Anxiety Disorder scale (GAD-7) | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  7-items self-report instrument for severity of anxiety symptoms, scores ranging from 0-21, higher scores indicating more severe anxiety
Work and Social Adjustment Scale (WSAS) | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  5-item self-report instrument for impairment of functioning, scores ranging from 0-40, higher scores indicating more impairment in functioning
Mental Health Quality of Life questionnaire (MHQoL) | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  7-item self report instrument for quality of life measure for use in people with mental health problems, scores ranging from 0-21, higher scores indicating higher quality of life, and MHQoL-VAS visual scale ranging from 0 (worst imaginable psychological wellbeing) to 10 (best imaginable psychological wellbeing)
Dysfunctional beliefs and attitudes about sleep (DBAS-10) | Baseline (T0), 3 weeks after baseline (T1), 6 weeks after baseline (T2)
  10-item abbreviated measure for dysfunctional beliefs and attitudes about sleep, scored on a scale from 0 (strongly disagree) to 10 (strongly agree)
Pre-Sleep Arousal Scale (PSAS) | Baseline (T0), 3 weeks after baseline (T1), 6 weeks after baseline (T2)
  16-item self report instrument for pre-sleep arousal, 5-point Likert Scale, higher scores reflecting more arousal
Academic performance | Baseline (T0), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  Students will be asked about the grade of their last exam (Scale 1-10), the average grade of the past semester (Scale 1-10), whether they failed any exams in the past semester (Yes/No), and their study progression in the past semester in terms of ECTS achieved (30 ECTS per semester, Yes/No)

OTHER OUTCOMES:
Adherence - Total number of completed modules | Through study completion, an average of 18 weeks
  Measures though Log Data
Adherence - Time spent in the platform (in minutes) | Through study completion, an average of 18 weeks
  Measures though Log Data
Adherence - Number of logins (total amount) | Through study completion, an average of 18 weeks
  Measures though Log Data
Adverse events | Mid-treatment (T1), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  1) falling accidents, 2) traffic accidents, or 3) any other accidents related to fatigue or sleepiness, and its consequences
Stressful life events questionnaire | Baseline (T0), 3 weeks after baseline (T1), 6 weeks after baseline (T2), and 18 weeks after baseline (T3)
  2 item questionnaire about whether participants experienced life-threatening or serious accident/ illness, death of someone close, physical/sexual violence or abuse or other incidents, and the consequences thereof

CONTACTS AND LOCATIONS:
Overall Officials: Niki Antypa, Dr., Principal Investigator — Leiden University
Locations (1):
- Leiden Univeristy, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pape LM, van Straten A, Struijs SY, Karch JD, Spinhoven P, Antypa N; Caring Universities Consortium. Effects of a Guided Digital Intervention on Sleep and Mental Health Outcomes in University Students - A Randomized Controlled Trial. Sleep. 2025 Nov 25:zsaf357. doi: 10.1093/sleep/zsaf357. Online ahead of print. PMID 41288591
- [Derived] Pape LM, van Straten A, Struijs SY, Spinhoven P, Antypa N. Effectiveness of a guided digital self-help intervention to improve sleep and the biological clock in university students - Study protocol for a randomized controlled trial. Internet Interv. 2024 Aug 2;37:100763. doi: 10.1016/j.invent.2024.100763. eCollection 2024 Sep. PMID 39224668